CLINICAL TRIAL: NCT01506362
Title: An Open-Label Study to Evaluate the Efficacy, Pharmacodynamics, Safety and Tolerability of Oral BL-7040 in Patients With Moderately Active Ulcerative Colitis
Brief Title: Efficacy, Pharmacodynamics, Safety and Tolerability of Oral BL-7040 in Patients With Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-7040.01
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; IBD
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A synthetic oligonucleotide for treatment of IBD. (Experimental): BL-7040 is an orally available new chemical entity for the treatment of IBD. BL-7040 is a synthetic oligonucleotide with dual activity on both the nervous and immune systems.
  Interventions: Drug: BL-7040

INTERVENTIONS:
Drug: BL-7040 — BL-7040 is an orally available new chemical entity for the treatment of IBD. BL-7040 is a synthetic oligonucleotide with dual activity on both the nervous and immune systems.
  Study duration can last up to 8 weeks, including up to 9 days in the screening period, up to 5 weeks of treatment with BL-7040, and up to 2 weeks for follow up.
  BL-7040 12 mg QD for 19-21 days followed by BL-7040 40 mg QD for 14 days.

SUMMARY:
The objective of the proposed study is to determine whether BL-7040 demonstrates clinical efficacy in patients with inflammatory bowel disease (IBD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 70.
2. Moderately active ulcerative colitis as defined by Mayo score of ≥ 5 and ≤ 9 within 9 days of first day of study treatment.
3. Diagnosis of ulcerative colitis ≥ 3 months prior to study entry.
4. Endoscopic sub-score of ≥ 2 and rectal bleeding sub-score of ≥ 1 on the Mayo score and endoscopic evidence of disease activity a minimum of 20 cm from the anal verge, determined within 9 days of first day of study treatment.
5. Female patients must have a negative serum pregnancy test at screening and be willing and able to use a medically acceptable method of birth control or declare that they are abstaining from sexual intercourse, from the screening visit through the study termination visit or be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal. Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
6. Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment

Exclusion Criteria:

1. Diagnosis of indeterminate colitis or clinical findings suggestive of Crohn's disease.
2. Subjects with ulcerative proctitis.
3. A diagnosis of ischemic colitis, fulminant colitis or toxic megacolon.
4. Evidence of bowel infection.
5. Body temperature ≥ 38°C at screening.
6. Evidence of abdominal abscess at the initial screening visit.
7. Extensive colonic resection, subtotal or total colectomy.
8. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
9. Receiving non-permitted IBD therapies
10. History of or current peptic ulcer disease.
11. Pregnant or lactating women.
12. Chronic hepatitis B or C infection or HIV seropositivity.
13. Current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurological disease.
14. Drug or alcohol abuse (by history).
15. Patients participating in any other clinical trials.
16. Patients with inability to communicate well with the Investigators and staff (i.e., language problem, poor mental development or impaired cerebral function).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Fishman, MD, Principal Investigator — Sourasky Medical Center; Eran Israeli, MD, Principal Investigator — Hadassah Medical Organization; Yehuda Chowers, MD, Principal Investigator — Rambam Health Care Campus; Eran Goldin, MD, Principal Investigator — Shaare Zedek Medical Center; Alex Fisch, MD, Principal Investigator — Soroka University Medical Center
Locations (5):
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah medical center, Jerusalem
  - Shaare Zedek Medical center, Jerusalem
  - Sourasky Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- A Synthetic Oligonucleotide for Treatment of IBD.: BL-7040 is an orally available new chemical entity for the treatment of IBD. BL-7040 is a synthetic oligonucleotide with dual activity on both the nervous and immune systems.
  Study duration can last up to 8 weeks, including up to 9 days in the screening period, up to 5 weeks of treatment with BL-7040, and up to 2 weeks for follow up.
  BL-7040 12 mg QD for 19-21 days followed by BL-7040 40 mg QD for 14 days.
Period: Overall Study
Arm/Group | A Synthetic Oligonucleotide for Treatment of IBD.
Started | 22
Completed | 16
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- A Synthetic Oligonucleotide for Treatment of IBD.: BL-7040 is an orally available new chemical entity for the treatment of IBD. BL-7040 is a synthetic oligonucleotide with dual activity on both the nervous and immune systems.
  BL-7040: BL-7040 is an orally available new chemical entity for the treatment of IBD. BL-7040 is a synthetic oligonucleotide with dual activity on both the nervous and immune systems.
  Study duration can last up to 8 weeks, including up to 9 days in the screening period, up to 5 weeks of treatment with BL-7040, and up to 2 weeks for follow up.
  BL-7040 12 mg QD for 19-21 days followed by BL-7040 40 mg QD for 14 days.
Arm/Group | A Synthetic Oligonucleotide for Treatment of IBD.
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (13.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants]
  Israel | 22

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who After Study Completion Achieve Clinical Response Defined by at Least a 3point Decrease & 30% Reduction From Baseline in Mayo Score Plus ≥ 1 Point Decrease in Rectal Bleeding Sub-score or Absolute Rectal Bleeding Subscore of ≤ 1
Description: Mayo score assesses stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment. It is assessed according to the following parameters:
  Stool frequency (subscore 0-3) 0: Normal number of stools for patient
  1. 1 to 2 stools per day more than normal
  2. 3 to 4 stools more than normal
  3. > or = to 5 stools more than normal
  Rectal bleeding (subscore 0-3) 0: No blood seen
  1. Streaks of blood with stool less than half the time
  2. Obvious blood with stool most of the time
  3. Blood alone passes
  Endoscopic findings (subscore 0-3) 0: Normal or inactive disease
  1 Mild Disease (erythema, decreased vascular pattern, mild friability) 2: Moderate Disease (marked erythema, lack of vascular pattern, friability erosions) 3: Severe Disease (spontaneous bleeding, ulceration)
  Physician's Global Assessment (subscore 0-3) 0: Normal
  1. Mild disease
  2. Moderate disease
  3. Severe disease
Time Frame: From Baseline to day 34 (end of treatment period)
Measure: Number; unit: participants
Arm/Group | A Synthetic Oligonucleotide for Treatment of IBD.
Number analyzed (Participants) | 22
participants | 8

2. Secondary Outcome: Proportion of Patients With Mucosal Healing After Completion of Study Treatment Defined as Reduction in Endoscopy Subscore of ≥ 1 From Baseline & an Absolute Endoscopy Subscore of ≤ 1 Assessed by Flexible Sigmoidoscopy.
Time Frame: 5 weeks following first administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | A Synthetic Oligonucleotide for Treatment of IBD.
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Synthetic Oligonucleotide for Treatment of IBD. (N=22)
hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Synthetic Oligonucleotide for Treatment of IBD. (N=22)
Exacerbation of ulcerative colitis (Gastrointestinal disorders) | 4 (4)
Influenza-like illness (General disorders) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No